CLINICAL TRIAL: NCT00887835
Title: A Post-Market Study of Transfacet Lumbar Spine Fixation and Fusion Utilizing the PERPOS™ PLS System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Interventional Spine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLS-007-FUS
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Lumbar Facet Disease
Keywords: PERPOS fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PERPOS™ PLS (Experimental): Minimally invasive transfacet fixation with PERPOS™ PLS as an aid to fusion
  Interventions: Device: PERPOS™ PLS

INTERVENTIONS:
Device: PERPOS™ PLS — To stabilize the spine as an aid to fusion through bilateral immobilization of the facet joints.

SUMMARY:
The purpose of this study is to utilize the PERPOS™ PLS System for transfacet lumbar spine fixation to evaluate its effect on patients' level of pain, procedural complications and functional status.

DETAILED DESCRIPTION:
The PERPOS™ PLS System involves a minimally invasive, percutaneous implant procedure via a small incision.

The PERPOS™ PLS is intended for lumbar bilateral facet fixation, with or without bone graft, at single or multiple levels from L1 to S1.

ELIGIBILITY:
Inclusion Criteria:

* Females and males between 18 and 85
* Must have lumbar facet disease confirmed by:

  1. Documented pain relief with controlled lumbar facet block using local anesthetic or steroid administration; AND
  2. MRI or CT scan, with or without bone scan, obtained within 3 months of enrollment, confirming arthritic facet joints OR, must have lumbar facet disease (as confirmed above) and are contra-indicated for steroid injections, or non-compliant with conservative pain management treatments, or wish to avoid the side-effects of steroids or prescriptive pain medication treatment
* Must score at least 4 on a 10-point Visual Analog Scale (VAS) for back pain
* Must score at least 40% on the Oswestry Disability Index.
* Must have less than 50% disc height loss
* Must have no greater than Grade I spondylolisthesis demonstrated on flexion and extension lumbar radiographs taken within 2 months of enrollment
* Willing and able to comply with the requirements of the protocol including follow-up requirements
* Willing and able to sign a study specific informed consent.

Exclusion Criteria:

* Are within the first two PERPOS PLS System utilization experience of the investigator
* Have severe facet degeneration, radiographic findings of severe facet joint disease, degeneration of misshapen facet(s) or structural anomalies at the target fusion level that would preclude proper placement of the BONE-LOK Implant.
* Have evidenced malingering behavior related to workman's compensation claims
* Have had any significant prior intervention (greater than an injection) in the facet joint to be treated, or within two (2) levels above or two (2) levels below the facet joint to be treated
* Have had prior instrumentation of involved vertebrae at any time
* Have osteoporotic bone at the lumbar spine level to be treated based on the SCORE (Simple Calculated Osteoporosis Risk Estimation) screening questionnaire, (or a DEXA bone density measured T score <-1.0.).
* Have scoliosis with lateral angulation >20 degrees
* Have an active malignancy: A subject with a history of any invasive malignancy (except non-melanoma skin cancer), unless s/he has been treated with curative intent and there have been no clinical signs or symptoms of malignancy for at least 5 years.
* Have a cyst in the canal associated with the facet
* Have neurologic deficit bowel or bladder dysfunction
* Have spinal canal or neural foramen compromise
* Have an infection (local or systemic)
* Have myelopathy
* Have abnormal coagulation time
* Have been or will be on anticoagulation therapy within 10 days of the study procedure
* Have radiculopathy
* Have cord compression or canal compromise requiring surgery for decompression
* Have disabling back pain secondary to another cause
* Have COPD that poses anesthesia risk
* Have severe cardiopulmonary deficiencies
* Have narcotic dependence or >90 days of narcotic pain medications
* Are morbidly obese (BMI >40)
* Have uncontrolled diabetes
* Have known allergies to implant materials, e.g., titanium.
* Are currently pregnant or lactating or considering becoming pregnant during the follow-up period
* Have been involved in an investigational drug or device study within the previous 30 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index and Visual Analogue Scale | 1 year